CLINICAL TRIAL: NCT04894968
Title: Identifying Predictors for the Development and Uphold of Heart Failure With Preserved Ejection Fraction
Brief Title: Prediction of the Development of Heart Failure With Preserved Ejection Fraction
Acronym: PREDICT-HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT-HFpEFv1
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure with preserved ejection fraction; Heart failure; Adiposity; Inflammation
MeSH Terms: conditions — Heart Failure; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of the presence of heart failure with preserved ejection fraction, according to guideline recommendations from the European Society of Cardiology 2016 — Patient will be screened for the presence of heart failure with preserved ejection fraction, according to guideline recommendations from the European Society of Cardiology 2016.
  This requires patients to fulfill all of the four criteria listed below:
  1. Symptoms of heart failure (e.g. dyspnea on extertion)
  2. Preserved ejection fraction (Left ventricular ejection fraction ≥50%
  3. NT-proBNP ≥125 pg/mL
  4. Echocardiographic signs for structural heart disease or diastolic dysfunction (at least one of the criteria below)
     * Left atrial volume index >34 mL/m²
     * Left ventricular mass index ≥115 g/m² for males or ≥95 g/m² for females
     * E/e' ≥13
     * Septal e' <9 cm/s

SUMMARY:
The ultimate goal of the PREDICT-HFpEF study is to identify and unravel predictors for the development of heart failure with preserved ejection fraction (HFpEF) in a cohort at increased cardiovascular risk. Patients that were initially included in another prospective cohort study (LIFE-Heart study) and did not show evident heart failure at that timepoint, will be followed-up approximately 7-years after their initial inclusion in the LIFE-Heart study. Patients will be screened for the development of HFpEF and characterized with thorough clinical as well as laboratory assessment. Patients will be classified according to the presence of absence of heart failure and predictors for the development will be identified by using measurements taken at their initial inclusion in the LIFE-Heart study.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is associated with severe morbidtiy and mortality. Yet, little is known about factors leading to the development of HFpEF investigated in a longitudinal fashion. The PREDICT-HFpEF study aims to adress this open question. Patients that were initially included in a large cohort study (LIFE-Heart study) approximately 7-years ago, that underwent thorough clinical, laboratory and echocardiographic assessment, and did not show evidence of heart failure at the present time point will be included in the current study.

Patients will be screened for the development of HFpEF or other forms of heart failure (e.g. heart failure with reduced ejection fraction) and will again undergo thorough clinical, laboratory and echocardiographic assessment. Initially measured biomarkers (including clinical data, lab-charts, ECG recordings and echocardiography) will be used to predict the development of HFpEF in this cohort at cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* At timepoint of inclusion in the LIFE-Heart study normal left ventricular ejection fraction (≥ 50%)
* At timepoint of inclusion in the LIFE-Heart study normal NT-proBNP (< 125 ng/l)

Exclusion Criteria:

* At timepoint of inclusion in the LIFE-Heart study acute coronary syndrom

  1. Troponine elevation above 14 pg/ml as well as coronary intervention, or isolated troponine elevation above 50 pg/ml in the absence of a coronary intervention
  2. No troponine elevation but coronary intervention
  3. Creatine kinase > 0.41 µmol/l*s and Creatine kinase to Creatine kinase-MB ration >6% or Creatine kinase-MB > 0.82 µmol/l*s
* At timepoint of inclusion in the LIFE-Heart study missing data on left ventricular ejection fraction
* At timepoint of inclusion in the LIFE-Heart study missing NT-proBNP measurement
* At timepoint of inclusion in the LIFE-Heart study missing data on echocardiographic diastolic function and structural alterations of the left ventricle
* At timepoint of inclusion in the LIFE-Heart study relevant valvular heart disease (including relevant aortic stenosis, mitral- and/or tricuspid regurgitation, congenital heart disease, mitral stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without evident heart failure with preserved ejection fraction that were included in the prospective cohort study: LIFE-Heart
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Heart failure with preserved ejection | At timepoint of inclusion
  Presence of heart failure with preserved ejection fraction according to the European Society of Cardiology 2016 criteria

SECONDARY OUTCOMES:
Occurence of major adverse cardiovascular events | 24-months after study inclusion
  Patients will be followed-up after their inclusion in the PREDICT-HFpEF study for the occurence of major adverse cardiovascular events using regular telephone interviews.
Changes in vascular status | At timepoint of inclusion
  Patients vascular status will be screened at study inclusion (e.g. intima media thickness) and will be set in relation to initially assessed vascular status at their initial inclusion in the LIFE-Heart study
Changes in organ function | At timepoint of inclusion
  Patients liver, as well as renal function as assessed by laboratory status will be screened at study inclusion (e.g. creatinine, bilirubine, Gamma-glutamyltransferase) and will be set in relation to initially assessed vascular status at their initial inclusion in the LIFE-Heart study
All-cause death | Yearly, after study enrollment up to ten years
  Patients will be screened on a yearly basis for the occurence of all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig at Leipzig University, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rommel KP, von Roeder M, Latuscynski K, Oberueck C, Blazek S, Fengler K, Besler C, Sandri M, Lucke C, Gutberlet M, Linke A, Schuler G, Lurz P. Extracellular Volume Fraction for Characterization of Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2016 Apr 19;67(15):1815-1825. doi: 10.1016/j.jacc.2016.02.018. PMID 27081022
- [Background] Rommel KP, von Roeder M, Oberueck C, Latuscynski K, Besler C, Blazek S, Stiermaier T, Fengler K, Adams V, Sandri M, Linke A, Schuler G, Thiele H, Lurz P. Load-Independent Systolic and Diastolic Right Ventricular Function in Heart Failure With Preserved Ejection Fraction as Assessed by Resting and Handgrip Exercise Pressure-Volume Loops. Circ Heart Fail. 2018 Feb;11(2):e004121. doi: 10.1161/CIRCHEARTFAILURE.117.004121. PMID 29449367